CLINICAL TRIAL: NCT07004257
Title: ButOx Human Trial: An Open Label Prospective Cohort Study to Investigate the Effect of Tributyrin (Butyrate Precursor Molecule) Supplementation on Markers of Calcium Oxalate Nephrolithiasis
Acronym: ButOx
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Ben Chew, MD, Associate Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H25-00547
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Urolithiasis
Keywords: Urolithiasis; Kidney Stones; Urinary Caliculi
MeSH Terms: conditions — Urolithiasis; Kidney Calculi | interventions — tributyrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tributyrin (Experimental): tributyrin (875 mg, BID)
  Interventions: Dietary Supplement: tributyrin

INTERVENTIONS:
Dietary Supplement: tributyrin — tributyrin (875 mg, BID)

SUMMARY:
Kidney stone disease (KSD) is a condition where there are crystal deposits in the kidney. The gut microbiome is a community of gut bacteria which can produce substances such as short chain fatty acids (SCFAs). Individuals with KSD have a different gut microbiome composition and lower amounts of these SCFAs compared to healthy individuals. Tributyrin is a supplement which can increase levels of SCFAs. Our data from animal studies indicate that tributyrin supplementation may be able to reduce kidney stone formation. This pilot clinical trial will test if tributyrin supplementation helps in prevention or treatment of those with KSD.

DETAILED DESCRIPTION:
Purpose

The objective of this pilot study is to understand how the butyrate prodrug, tributyrin (875 mg, BID) influences urine and stool parameters of kidney stone disease.

Hypothesis

The hypothesis of this study is that the tributyrin is able to reduce levels of markers related to stone formation. There has been no study to date which investigates the potential for tributyrin or other butyrate supplements in relationship to these markers of kidney stone disease. Through this pilot study we plan to capture sufficient data in a small group of individuals to understand the clinical implications for tributyrin supplementation.

Justification

While there are a variety of options for treating kidney stones, preventative measures are lacking and largely include a variety of lifestyle changes. A dysbiotic gut microbiome has been implicated in kidney stone disease for the past 20-years, however we have yet to develop effective therapeutics which target the gut microbiome. Experiments in our lab indicate that tributyrin significantly reduces kidney crystal deposits in a murine model of kidney stone disease. As such it is important to understand if tributyrin modulates levels of urine and stool parameters related to kidney stone disease.

Objectives

The objectives of this study are to:

1. Investigate tributyrin supplementation to increase butyrate levels (stool, blood) in a population with a history of calcium oxalate nephrolithiasis
2. Understand how tributyrin supplementation influences measures related to stone formation

Study Endpoints

The primary endpoint of this study is change in serum butyrate levels when comparing baseline (pre-tributyrin) and endpoint (post-tributyrin) levels.

Secondary endpoints include:

1. Changes in urine oxalate levels
2. Changes in stool oxalate levels
3. Changes in stool butyrate levels
4. Changes in urinary chemical levels (citrate, calcium, phosphate, uric acid, creatinine, and pH)
5. Changes in urinary inflammatory markers (IL-6, IL-8, IL-10, and IL-18)
6. Changes in urinary markers of oxidative stress (8-OHdG)
7. Changes in microbiome composition
8. Measurement of nutrient intake using ASA24® dietary assessment tool (oxalate, calcium, dietary fibre, and water intake)
9. Measurement of crystalluria

Statistical Analysis

For our pilot trial we plan to recruit 10 subjects and use a within-subjects design. Since this is a pilot study, we will use the results for power calculations to understand an appropriate sample size for a larger study. Data collected from the biological samples will be analyzed with the paired-samples t-test. Due to the novelty of this research in humans, we will run covariate analyses on our pilot data to determine which variables may be confounding, but we expect to include variables such as sex, age, number of previous kidney stones, and dietary habits. Microbiome data will be analyzed in our sequencing facility at The Stone Centre. The ASA24® dietary assessment data will be analyzed using the ASA24® Researcher Website and consumption of oxalate, calcium, and hydration status will be used for dietary habit analysis.

If we see a significant elevation (p<0.05) in serum butyrate levels, accompanied by changes in oxalate excretion (indicated by stool, serum, and urine oxalate levels) and changes in urine biomarkers in individuals taking the tributyrin supplement this trial will be successful, and be continued in follow-up experiments.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years.
2. History of nephrolithiasis, diagnosed with a kidney stone containing >80% calcium (from stone analysis of spontaneously passed or surgically removed kidney stone) within the past 3 years
3. Written informed consent

Exclusion Criteria:

1. Pregnant or lactating females
2. Pharmacological therapy for stone disease over the last moth (aside from an increase in water intake)
3. Antibiotic use in the last 3 months prior to the start of study procedures (start of baseline period)
4. Subjects with comorbid conditions which may influence the microbiome or increase the risk of nephrolithiasis (inflammatory bowel diseases, bariatric surgery, active malignancy, celiac disease, cystic fibrosis, diabetes mellitus, urinary tract obstruction, renal tubular acidosis)
5. Chronic intestinal diseases, or bowel resection surgeries
6. Inability to provide informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Tributytin Levels | 28 Days
  change in serum butyrate levels when comparing baseline (pre-tributyrin) and endpoint (post-tributyrin) levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No